CLINICAL TRIAL: NCT01119209
Title: Postoperative Analgesia With Local Infiltration After Hip Fracture Of Intertrochanteric Type
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Rune Dueholm Bech, MD, Odense University Hospital, DK-5000 Odense C, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S-VF-20060072 - trochanteric
Record Dates: First submitted 2010-05-04; First posted 2010-05-07 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Hip Fracture of Intertrochanteric Type
Keywords: Hip fracture; intertrochanteric
MeSH Terms: conditions — Hip Fractures | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine (Active Comparator)
  Interventions: Drug: Ropivacaine; Drug: Saline
- Saline (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ropivacaine — Approved by the Danish Medicines Agency
  Arms: Ropivacaine
Drug: Saline — Approved by the Danish Medicines Agency

SUMMARY:
Reducing pain is an essential factor for early mobilization after osteosynthesis of intertrochanteric fractures. Systemic opioids have side effects that might obstruct mobilization and induce delirium and nausea. The investigators hypothesized that wound infiltration results in reduction in systemic opioid usage and pain relief without side effects.

ELIGIBILITY:
Inclusion Criteria:

* Intertrochanteric hip fracture
* Fracture due to low energy trauma
* Ability to understand danish and give informed consent
* Ability to walk before trauma
* Indication for osteosynthesis

  •≥ 8 in OMC (Orientation-Memory-Concentration) test with a possible maximum of 28 points
* Informed consent

Exclusion Criteria:

* Drug or medical abuse
* Drug intolerance
* Pathological fractures
* Inflammatory arthritis
* Patient included in the study with the contralateral hip

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2008-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Consumption of opioids | 5 days postoperatively

SECONDARY OUTCOMES:
Pain | 5 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Soren Overgaard, MD, DmSc, Study Chair — Odense University Hospital, DK-5000 Odense C, Denmark; Rune Dueholm Bech, MD, Principal Investigator — Odense University Hospital, DK-5000 Odense C, Denmark
Locations (1):
- Odense University Hospital, Odense, DK, Denmark

REFERENCES:
- [Derived] Bech RD, Ovesen O, Lauritsen J, Emmeluth C, Lindholm P, Overgaard S. Local Anesthetic Wound Infiltration after Osteosynthesis of Extracapsular Hip Fracture Does Not Reduce Pain or Opioid Requirements: A Randomized, Placebo-Controlled, Double-Blind Clinical Trial in 49 Patients. Pain Res Manag. 2018 Nov 13;2018:6398424. doi: 10.1155/2018/6398424. eCollection 2018. PMID 30538796